CLINICAL TRIAL: NCT03548142
Title: Palliative and Hospice Care in Advanced Dementia: Experiences of Care Givers and Benefit of a Brochure Serving as a Decision-making Aid
Brief Title: Advanced Dementia and End-of-life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Bavarian State Ministry of Health and Care (Other Government); German Alzheimer Society (Other)
Responsible Party: Principal Investigator, Janine Diehl-Schmid, Clinical Professor, Principle Investigator, Technical University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: palliative study
Record Dates: First submitted 2017-11-13; First posted 2018-06-07 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Advanced Dementia
Keywords: Palliative Care; advanced dementia; life-prolonging treatment; patient will; advanced care planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: provision of relevant information — caregivers are provided with brochure that informs about end-of-life issues for persons with advanced dementia

SUMMARY:
Palliative and hospice care in advanced dementia: experiences of care givers and benefit of a brochure serving as a decision-making aid

Aims:

1. Designing a brochure serving as an information tool and decision-making aid used to answer questions concerning palliative and hospice care for care-givers of persons with advanced dementia.

   The brochure shall demonstrate the possibilities and offerings of palliative and hospice care and shall serve to inform about the advanced stages of dementia, the legal basic principles in decision making and ethical problems, treatment options and (palliative) treatment goals.
2. Survey of the palliative, palliative medical and hospice care of persons with advanced dementia in ambulatory settings, as well as in residential geriatric care and the experiences of the care-givers.

   By examining persons with dementia and inspecting the care documents and where applicable the medical files it is to be evaluated:
   * which procedures of palliative and hospice care are practically implemented in ambulatory care and in residential geriatric care,
   * which symptoms the persons with dementia suffer from and how those symptoms are (or are not) treated,
   * to what extend caregivers are informed about relevant aspects
   * how caregivers assess care and which problems, needs and requests exist.
3. Piloting phase for the brochure. To test the comprehensibility and the acceptance of the brochure a study is planned. The caregivers are asked for their opinion whether the brochure is helpful. It is recorded if the reading of the brochure gets the caregivers to engage actively in the participative decision making process.

DETAILED DESCRIPTION:
Two visits at home or in the residential geriatric care at intervals of eight to twelve weeks are scheduled.

The following data is collected at enrollment:

* Informed consent of the caregiver and of the patient or rather the caregiver with powers of attorney
* Sociodemographic data (caregiver and person with dementia), e.g. age, sex, education, degree of relationship
* Interview of the caregiver using standardized
* Examination of the person with dementia, recording of the treatment and the care situation, cognitive status: Mini-Mental-Status-Test, severity of dementia: Clinical Dementia Rating Scale, performance in basic activities of daily living: Barthel-Index,communication competence, diagnosis, (palliative) medical and hospice care (including specialists in palliative care, specialists in hospice care, general practioners, domiciliary care services, Allgemeine Ambulante Palliativversorgung [AAPV], Spezielle Ambulante Palliativversorgung [SAPV], AAPV and SAPV both being a specific ambulatory palliative care of the statutory health insurance system in Germany, cognitive/neurological/physical symptoms, symptom Management including pharmacological and non-pharmacological treatment, interventions, existence and phrasing of advanced directives and durable power of attorney.

After enrollment the brochure is handed and explained to the caregivers and they are encouraged to read it. It is pointed out that they are contacted after two to three months to answer questions concerning comprehensibility, acceptance, practical consequences and to give a personnel review.

At study end after two to three months standardized interviews are conducted to gather information about comprehensibility and acceptance of the brochure, how it is reviewed by the caregivers and if the reading had direct consequences with regard to knowledge of the caregiver, communicating with nursing staff/physicians, decision making and implementing those decisions.

ELIGIBILITY:
Inclusion Criteria:

* Person with dementia + caregiver live in the Munich area
* Person with dementia lives in a nursing home or at home
* Person with dementia is in an advanced stage of the disease (moderate to severe dementia)
* Informed consent of the caregiver and the person with powers of attorney
* Caregiver is German-speaking and able to read

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Patients' Perceived Involvement in Care Scale | two to three months
  Involvement is expected, when caregiver at study end achieve one point more in the sum score (sum score maximum is eight points)

SECONDARY OUTCOMES:
family caregivers´satisfaction with care | Assessment A (inclusion/baseline, before reading the brochure) and Assessment B (after reading the brochure, two to three months after Assessment A)
  the adapted version of End of life in dementia-Satisfaction with Care, (SWC-EOLD)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Cognitive Disorders, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Lerman CE, Brody DS, Caputo GC, Smith DG, Lazaro CG, Wolfson HG. Patients' Perceived Involvement in Care Scale: relationship to attitudes about illness and medical care. J Gen Intern Med. 1990 Jan-Feb;5(1):29-33. doi: 10.1007/BF02602306. PMID 2299426
- [Background] Vohra JU, Brazil K, Hanna S, Abelson J. Family Perceptions of End-of-Life Care in long-term care facilities. J Palliat Care. 2004 Winter;20(4):297-302. PMID 15690832
- [Background] Biola H, Sloane PD, Williams CS, Daaleman TP, Williams SW, Zimmerman S. Physician communication with family caregivers of long-term care residents at the end of life. J Am Geriatr Soc. 2007 Jun;55(6):846-56. doi: 10.1111/j.1532-5415.2007.01179.x. PMID 17537084
- [Derived] Ryan RE, Connolly M, Bradford NK, Henderson S, Herbert A, Schonfeld L, Young J, Bothroyd JI, Henderson A. Interventions for interpersonal communication about end of life care between health practitioners and affected people. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD013116. doi: 10.1002/14651858.CD013116.pub2. PMID 35802350
- [Derived] Riedl L, Bertok M, Hartmann J, Fischer J, Rossmeier C, Dinkel A, Ortner M, Diehl-Schmid J. Development and testing of an informative guide about palliative care for family caregivers of people with advanced dementia. BMC Palliat Care. 2020 Mar 12;19(1):30. doi: 10.1186/s12904-020-0533-3. PMID 32164707
- See also: legal basis for AAPV and SAPV — https://www.gkv-spitzenverband.de/media/dokumente/krankenversicherung_1/hospiz_palliativversorgung/versorgungsplanung/Vereinbarung_nach_132g_Abs_3_SGBV_ueber_Inhalte_und_Anforderungen_der_gesundheitlichen_Versorgungsplanung.pdf
- See also: Preparation for decision making scale — https://decisionaid.ohri.ca/docs/develop/Tools/PrepDM.pdf